CLINICAL TRIAL: NCT06211452
Title: Comparison of Consolidation Strategies for Pediatric Patients With Acute Myeloid Leukemia - Results of the Randomized GATLA 8-LMA-P'07 Trial
Brief Title: Comparison of Consolidation Strategies for Pediatric Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GATLA 8-AML´07
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: AML; Pediatric AML
Keywords: AML; Pediatric AML; Randomization

STUDY DESIGN:
Intervention Model Description: It is a randomized model, the evaluation is based on event time (overall survival, event free survival, cumulative incidence relapse with treatment related mortality as competitive event). Comparator log rank test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: Conventional Consolidation (Active Comparator): Conventional consolidation (CONS) (active comparator) (6-thioguanine 60 mg/m2/d, on days 1 to 43 orally; prednisone 40 mg/m2/d, on days 1 to 28 orally; vincristine 1.5 mg/m2/d, on days 1, 8, 15, 22; idarubicin 7 mg/m2/d, on days 1, 8, 15, 22; cytarabine 75 mg/m2/d, on days 3-6, 10-13, 17-20, 24-27, 31-34, 38-41; intrathecal cytarabine on days 1, 15, 29, 43 [age-dependent dose]; cyclophosphamide 500 mg/m2/d, on days 29, 43)
  Interventions: Drug: ARM A: Active Comparator Drug
- ARM B: Blocks Therapy (Experimental): Block Therapy: AI block (randomized; cytarabine 500 mg/m2 as continuous infusion ×4 days and idarubicin 7 mg/m2 on days 3 and 5; intrathecal cytarabine on days 0 and 6), haM block (high-dose cytarabine 1 g/m2 every 12 hours for 3 days and mitoxantrone 10 mg/m2 on days 4 and 5, intrathecal cytarabine days 6 and 15)
  Interventions: Drug: ARM B: Blocks Therapy Drug

INTERVENTIONS:
Drug: ARM A: Active Comparator Drug — Consolidation 6-thioguanine 60 mg/m2/d, 1 to 43 po; prednisone 40 mg/m2/d, on days 1-28 orally; vincristine 1.5 mg/m2/d, days 1, 8, 15, 22; idarubicin 7 mg/m2/d, on days 1, 8, 15, 22; cytarabine 75 mg/m2/d, on days 3-6, 10-13, 17-20, 24-27, 31-34, 38-41; intrathecal cytarabine on days 1, 15, 29, 43; cyclophosphamide 500 mg/m2/d, days 29, 43.
  Arms: ARM A: Conventional Consolidation
Drug: ARM B: Blocks Therapy Drug — Blocks AI Cytarabine 500 mg/m2 as 24 infusion infusion x 4 d; Idarubicin 7 mg/m2 on days 3 and 5; Intrathecal cytarabine on days 0 and 6.
  haM Cytarabine 1 g/m2 every 12 hours for 3 days; Mitoxantrone 10 mg/m2 days 4 and 5; Intrathecal cytarabine days 6 and 15.
  Arms: ARM B: Blocks Therapy

SUMMARY:
GATLA 8-AML´07 trial is an multicenter phase III dose-optimization trial for the treatment of acute myeloid leukemias in children and adolescents. Patients are treated with a combination of intensive chemotherapy in combination with intrathecal-injection by CNS and haematopoietic stem cell transplantation.

The patients are stratified in a standard-group (SR) and a high risk-group (HR). SR was defined as FAB (French-American-British) M1/M2 with Auer rods; FAB M4eo or favorable cytogenetics [t(8;21)/AML1-ETO or inv(16) or t(16;16) and/or CBFB/MYH11)]; bone marrow blasts ≤5% on day 15. HR was defined as all others. SR patients were reclassified to the HR group if FLT3-ITD positive.

Based on the experience of the BFM group, it was decided to randomly evaluate whether the six-drug conventional consolidation stage can be replaced with the use of a consolidation based by block therapy on drugs of proven efficacy in AML with the aim of reducing residual disease, and the toxicity of this stage. Patients are randomized once the double induction is completed into those who will receive the conventional consolidation phase and those who will receive consolidation with the combination of high doses cytarabine and two different anthracyclines sequentially.

DETAILED DESCRIPTION:
All patients in the trial, whether standard risk (SR) or high risk (HR), receive 2 Induction courses: AIE and HAM and then are randomized to continue with the consolidation phase: a conventional consolidation (Arm A) with 6 drugs vs 2 blocks of chemotherapy that are incorporated in this protocol (AI and haM) (Arm B) and then an Intensification phase with high doses of cytarabine and etoposide. The difference between the SR and AR groups is that the former don't continue with the maintenance phase, while those in HR receive 1 year of Maintenance if they don't have a histoidentical family donor. SR patients according to cytogenetics and with < 5% blasts in the bone marrow on day 15, haven´t indication for TCHP in 1st CR. HR patients, with a histoidentical family donor, will be transplanted in the 1st. CR after the Consolidation phases or the AI and haM blocks, according to the treatment arm that corresponded to them by randomization

ELIGIBILITY:
Inclusion Criteria:

* De novo AML
* FAB M0-M7
* Primary myelosarcomas or acute mixed lineage leukemia / biphenotypic leukemia (predominantly myeloid).
* Written informed consent from patients, parents, or guardians was obtained at study entry in accordance with the Declaration of Helsinki

Exclusion Criteria:

* AML as secondary malignancy
* Children with Down's syndrome
* Accompanying diseases which do not allow therapy according to the protocol
* Pre-treatment for more than 14 days with another intensive induction therapy
* Patients with APL
* Patients with myelodysplasia
* Patients with blast crisis of Chronic Myeloid Leukemia
* Patients who die before starting treatment

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 258 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2015-03-15 (Actual); Study Completion 2015-12-21 (Actual)

PRIMARY OUTCOMES:
Determine if two-cycle consolidation reduced the cumulative incidence of relapse compared to conventional consolidation (CONS) among newly diagnosed pediatric patients with AML. | 72 months
  The GATLA 8-LMA-P'07 was a randomized trial including pediatric AML children in Argentina; the design was based on AML-BFM 98 with minor modifications.(10) Similar to AML-BFM 98, the trial compared two approaches to consolidation. The standard regimen was a 6-week consolidation phase (CONS), which was also used in AML-BFM 93 vs. the comparator regimen of two short chemotherapy cycles (two-cycle) with cytarabine plus idarubicin (AI) and high dose cytarabine plus mitoxantrone (haM). AML-BFM 98 previously demonstrated that haM was tolerable.10 We hypothesized that the two-cycle consolidation (two-cycle) would be associated with lower relapse rates related to dose intensification compared to the standard CONS approach.

SECONDARY OUTCOMES:
Evaluate Event-free survival (EFS) of pediatric patients with AML. | 72 months
  EFS was calculated from date of randomization to first event (death, resistant leukemia, relapse or secondary malignancy) or date of last follow-up.
Evaluate Overall Survival (OS) of pediatric patients with AML. | 72 months
  OS was also calculated from date of randomization to date of death or date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alcyra Fynn, Dr., Study Chair — Grupo Argentino de Tratamiento de la Leucemia Aguda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasche M, Zimmermann M, Borschel L, Bourquin JP, Dworzak M, Klingebiel T, Lehrnbecher T, Creutzig U, Klusmann JH, Reinhardt D. Successes and challenges in the treatment of pediatric acute myeloid leukemia: a retrospective analysis of the AML-BFM trials from 1987 to 2012. Leukemia. 2018 Oct;32(10):2167-2177. doi: 10.1038/s41375-018-0071-7. Epub 2018 Feb 22. PMID 29550834
- [Background] van Weelderen RE, Njuguna F, Klein K, Mostert S, Langat S, Vik TA, Olbara G, Kipng'etich M, Kaspers GJL. Outcomes of pediatric acute myeloid leukemia treatment in Western Kenya. Cancer Rep (Hoboken). 2022 Oct;5(10):e1576. doi: 10.1002/cnr2.1576. Epub 2021 Nov 22. PMID 34811958
- [Background] Zwaan CM, Kolb EA, Reinhardt D, Abrahamsson J, Adachi S, Aplenc R, De Bont ES, De Moerloose B, Dworzak M, Gibson BE, Hasle H, Leverger G, Locatelli F, Ragu C, Ribeiro RC, Rizzari C, Rubnitz JE, Smith OP, Sung L, Tomizawa D, van den Heuvel-Eibrink MM, Creutzig U, Kaspers GJ. Collaborative Efforts Driving Progress in Pediatric Acute Myeloid Leukemia. J Clin Oncol. 2015 Sep 20;33(27):2949-62. doi: 10.1200/JCO.2015.62.8289. Epub 2015 Aug 24. PMID 26304895
- [Background] Sung L, Aplenc R, Alonzo TA, Gerbing RB, Lehrnbecher T, Gamis AS. Effectiveness of supportive care measures to reduce infections in pediatric AML: a report from the Children's Oncology Group. Blood. 2013 May 2;121(18):3573-7. doi: 10.1182/blood-2013-01-476614. Epub 2013 Mar 7. PMID 23471307
- [Background] Fedorovsky JM, Cuervo LG, Luciani S. Pediatric cancer registries in Latin America: the case of Argentina's pediatric cancer registry. Rev Panam Salud Publica. 2017 Dec 5;41:e152. doi: 10.26633/RPSP.2017.152. eCollection 2017. PMID 31384271
- [Background] Howard SC, Ortiz R, Baez LF, Cabanas R, Barrantes J, Fu L, Pena A, Samudio A, Vizcaino M, Rodriguez-Galindo C, Barr RD, Conter V, Biondi A, Masera G; MISPHO Consortium Writing Committee. Protocol-based treatment for children with cancer in low income countries in Latin America: a report on the recent meetings of the Monza International School of Pediatric Hematology/Oncology (MISPHO)--part II. Pediatr Blood Cancer. 2007 Apr;48(4):486-90. doi: 10.1002/pbc.20989. PMID 16883600
- [Background] Gibson BE, Webb DK, Howman AJ, De Graaf SS, Harrison CJ, Wheatley K; United Kingdom Childhood Leukaemia Working Group and the Dutch Childhood Oncology Group. Results of a randomized trial in children with Acute Myeloid Leukaemia: medical research council AML12 trial. Br J Haematol. 2011 Nov;155(3):366-76. doi: 10.1111/j.1365-2141.2011.08851.x. Epub 2011 Sep 9. PMID 21902686
- [Background] Creutzig U, Zimmermann M, Bourquin JP, Dworzak MN, Fleischhack G, Graf N, Klingebiel T, Kremens B, Lehrnbecher T, von Neuhoff C, Ritter J, Sander A, Schrauder A, von Stackelberg A, Stary J, Reinhardt D. Randomized trial comparing liposomal daunorubicin with idarubicin as induction for pediatric acute myeloid leukemia: results from Study AML-BFM 2004. Blood. 2013 Jul 4;122(1):37-43. doi: 10.1182/blood-2013-02-484097. Epub 2013 May 23. PMID 23704089
- [Background] Fernandez HF, Sun Z, Yao X, Litzow MR, Luger SM, Paietta EM, Racevskis J, Dewald GW, Ketterling RP, Bennett JM, Rowe JM, Lazarus HM, Tallman MS. Anthracycline dose intensification in acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1249-59. doi: 10.1056/NEJMoa0904544. PMID 19776406
- [Background] Creutzig U, Zimmermann M, Lehrnbecher T, Graf N, Hermann J, Niemeyer CM, Reiter A, Ritter J, Dworzak M, Stary J, Reinhardt D. Less toxicity by optimizing chemotherapy, but not by addition of granulocyte colony-stimulating factor in children and adolescents with acute myeloid leukemia: results of AML-BFM 98. J Clin Oncol. 2006 Sep 20;24(27):4499-506. doi: 10.1200/JCO.2006.06.5037. PMID 16983120
- [Background] Creutzig U, Zimmermann M, Ritter J, Henze G, Graf N, Loffler H, Schellong G. Definition of a standard-risk group in children with AML. Br J Haematol. 1999 Mar;104(3):630-9. doi: 10.1046/j.1365-2141.1999.01304.x. PMID 10086807